CLINICAL TRIAL: NCT02503761
Title: Bolus Versus Prolonged Infusion of Meropenem in Newborn With Late Onset Sepsis: A Randomized Control Trial
Brief Title: Bolus Versus Prolonged Infusion of Meropenem in Newborn With Late Onset Sepsis
Acronym: BVPIMNBLOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abd Elazeez Attala Shabaan, Assistant professor, PhD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67890
Record Dates: First submitted 2015-06-09; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Late Onset Neonatal Sepsis
Keywords: meropenem; infusion; late-onset sepsis; newborn; management
MeSH Terms: conditions — Neonatal Sepsis | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion arm (Active Comparator): Infants will receive a loading dose of 20 mg/kg/dose every 8 hours for sepsis and 40 mg/kg/dose every 8 hours in meningitis and pseudomonas infection. Each dose will be infused over four hours.
  Interventions: Drug: Meropenem.
- Bolus group (Active Comparator): Infants will receive a loading dose of 20 mg/kg/dose every 8 hours for sepsis and 40 mg/kg/dose every 8 hours in meningitis and pseudomonas infection. Each dose will be infused over thirty minutes.
  Interventions: Drug: Meropenem.

INTERVENTIONS:
Drug: Meropenem. — Infants in both groups will receive a loading dose of 20 mg/kg/dose every 8 hours for sepsis and 40 mg/kg/dose every 8 hours in meningitis and pseudomonas infection

SUMMARY:
Newborns in the neonatal intensive care unit (NICU), especially premature ones with immature organ systems, frequently suffer nosocomial infections caused by microorganisms resistant to narrow-spectrum antibiotics like ampicillin and gentamicin and require introduction of new agents with a wider spectrum of activity.

Meropenem has activity against wide variety of Gram-negative and Gram-positive bacteria. It is well tolerated by children and neonates, including preterm babies, and allowing monotherapy instead of combined therapy.

Severe neonatal infections with increasing antibiotic resistance are major problems affecting morbidity and mortality in the NICU. Few number of new antibacterial agents entering the clinic and new agents for multi-drug resistant Gram-negative bacteria will unlikely be available in the near future.

DETAILED DESCRIPTION:
More research into existing antibiotics with novel mechanisms of action are required to combat the increased resistance and decreased development of antibiotics. Efforts were exerted to maximize antibiotic efficacy by optimal dosing based on pharmacodynamic and pharmacokinetic properties of antibiotics.

Meropenem is administered mostly via a 30-min infusion, as some data indicate rapid degradation after reconstitution. Dose recommendations from two pediatric studies using Monte Carlo simulation have emphasized that a 4-h infusion may be needed if microorganisms showed increased minimal inhibitory concentrations (MICs), more specifically, for Pseudomonas aeruginosa. A prolonged-infusion strategy has not been tested in neonates, although some data suggest that extremely small infusion volumes may significantly affect the drug amount actually delivered.

Aim of work:

The objective of our study is to compare the clinical and bacteriological efficacy of conventional intermittent dosing of meropenem to the prolonged infusions in critically-ill neonates, with a proactive focus on reducing ventilator days in ventilated patients, length of stay in NICU, and neonatal mortality.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the neonatal care unit (NCU) who suffer from late onset sepsis (LOS) at admission or during their NICU stay and receive meropenem for at least four days

Exclusion Criteria:

* Acute or chronic renal failure
* Hypersensitivity or allergy to meropenem

Ages: 3 Days to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | 15-28 days from Meropenem treatment
  * Success is defined as complete or partial resolution of leukocytosis, temperature, and clinical signs and symptoms of infection.
  * Failure consists of persistence or progression of signs and symptoms of infection, development of new clinical findings consistent with active infection, or death from infection.
Microbiological outcome | 7-21 days from Meropenem treatment
  * Success is defined as eradication of infection or colonization which means detection of a new pathogen from the site of infection during meropenem therapy and no new antibiotic is indicated
  * Failure is defined as persistence of infection and superinfection which means detection of a new pathogen from the site of infection during meropenem therapy and new antibiotic is indicated.

SECONDARY OUTCOMES:
Meropenem-related length of mechanical ventilation | 0-31 days from Meropenem treatment
  The number of mechanical ventilation days from the start of meropenem administration
Meropenem-related length of NICU stay | 10 weeks from Meropenem treatment
  The number of days from the beginning of meropenem therapy to discharge from NICU
NICU mortality | 12 weeks from time of admission
  Death before discharge
Duration of meropenem treatment | 3-28 days
  Total days of meropenem treatment
Clinical side effects of meropenem treatment | 3-28 days from meropenem treatment
  Safety of meropenem therapy will be evaluated by clinical symptoms (diarrhea, rash, vomiting and seizures).
Laboratory derangement related to meropenem treatment | 3-28 days from meropenem treatment
  Assessment of laboratory parameters and their changes during meropenem therapy (transaminases, alkaline phosphatase, bilirubin).

REFERENCES:
- [Derived] Shabaan AE, Nour I, Elsayed Eldegla H, Nasef N, Shouman B, Abdel-Hady H. Conventional Versus Prolonged Infusion of Meropenem in Neonates With Gram-negative Late-onset Sepsis: A Randomized Controlled Trial. Pediatr Infect Dis J. 2017 Apr;36(4):358-363. doi: 10.1097/INF.0000000000001445. PMID 27918382